CLINICAL TRIAL: NCT01641159
Title: A Randomized Controlled Evaluation of Buspirone for Relapse-Prevention in Adults With Cocaine Dependence (BRAC)
Brief Title: Study of Buspirone for Relapse-Prevention in Adults With Cocaine Dependence
Acronym: BRAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Theresa Winhusen, Associate Professor, Department of Psychiatry and Behavioral Neuroscience; CinARC Director, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTN-0052; U10DA013732 (NIH)
Record Dates: First submitted 2012-07-10; First posted 2012-07-16 (Estimated); Results first posted 2014-12-17 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2014-12

CONDITIONS: Cocaine Dependence
Keywords: Cocaine; Crack; Buspirone; Relapse Prevention
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Buspirone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Buspirone plus TAU (Active Comparator): Buspirone titrated to 60 mg/day for the 15-week active study
  Interventions: Drug: Buspirone
- Placebo plus TAU (Placebo Comparator): Placebo taken daily for the 15-week active study
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Buspirone — Study participants will be randomly assigned to receive either buspirone or matching placebo. Following dose escalation, the target at study day 10 is to achieve the highest tolerated dose not exceeding 60 mg. Participants who are unable to reach the 60 mg dose or who need to be reduced from 60 mg due to tolerability will be maintained on 15 mg, 30 mg, or 45 mg, whichever is the highest dose tolerated.
  Other Names: Buspirone hydrochloride, Buspar
  Arms: Buspirone plus TAU
Drug: Placebo — Study participants will be randomly assigned to receive either buspirone or matching placebo. Placebo tablets will be identical in color and size to the buspirone tablets.
  Other Names: Matched placebo
  Arms: Placebo plus TAU

SUMMARY:
The purpose of this study is to evaluate whether or not buspirone is effective in preventing relapse in cocaine-dependent adults in inpatient/residential treatment who are planning to enter outpatient treatment upon inpatient/residential discharge.

DETAILED DESCRIPTION:
The primary objective is to evaluate the efficacy of buspirone, relative to placebo, in preventing relapse in cocaine-dependent adults in inpatient/residential treatment who are planning to enter outpatient treatment upon inpatient/residential discharge. Secondary objectives include evaluating the impact of buspirone, relative to placebo, on other drug-abuse outcomes and on factors that may mediate buspirone's efficacy as a relapse-prevention treatment.

ELIGIBILITY:
Inclusion Criteria:

1. be 18 years of age or older
2. be able to understand the study, and having understood, provide written informed consent in English
3. meet DSM-IV-TR diagnostic criteria for current (within the last 12 months) dependence for cocaine, must self-report having used crack cocaine a minimum of four times in the 28 days prior to inpatient/residential admission, and must report that their typical pattern of use is at least once a week
4. have a willingness to comply with all study procedures and medication instructions
5. be enrolled in an inpatient/residential program at a participating CTP, scheduled to be in inpatient/residential treatment for 12-19 days when randomized, and planning to enroll in local outpatient treatment through the end of the active treatment phase (i.e., study week 15)
6. if female and of child bearing potential, agree to use one of the following methods of birth control:

   * oral contraceptives
   * contraceptive patch
   * barrier (diaphragm or condom)
   * intrauterine contraceptive system
   * levonorgestrel implant
   * medroxyprogesterone acetate contraceptive injection
   * complete abstinence from sexual intercourse
   * hormonal vaginal contraceptive ring

Exclusion Criteria:

1. meet DSM-IV-TR diagnostic criteria for current (within the last 12 months) opioid dependence
2. have a medical or psychiatric condition that, in the judgment of the study physician, would make study participation unsafe or which would make treatment compliance difficult. Medical conditions that may compromise participant safety or study conduct include, but are not limited to:

   * AIDS according to the current CDC criteria for AIDS
   * liver function tests greater than 3X upper limit of normal
   * serum creatinine greater than 2 mg/dL
3. have a psychiatric disorder requiring continued treatment with a psychotropic medication
4. have a known or suspected hypersensitivity to buspirone
5. be pregnant or breastfeeding
6. have used any of the following medications within 14 days of randomization: monoamine oxidase (MAO) inhibitors such as phenelzine (Nardil), selegiline (Eldepryl), isocarboxazid (Marplan), or tranylcypromine (Parnate)
7. be taking any medications which, in the judgment of the study physician, may produce interactions with buspirone that are sufficiently dangerous so as to exclude the patient from participating in the study. Alternatively, the study physician, in consultation with the patient and his or her physician, may elect to withdraw the patient from the problem medications before randomization. Some of the possible interactions are discussed in section 8.8.
8. be anyone who, in the judgment of the investigator, would not be expected to complete the study protocol (e.g., due to relocation from the clinic area, probable incarceration, etc.)
9. be a significant suicidal/homicidal risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Winhusen, PhD, Principal Investigator — University of Cincinnati, CTN Ohio Valley Node
Locations (6):
- United States (6):
  - Gateway Community Services, Jacksonville, Florida
  - Maryhaven Inc, Columbus, Ohio
  - Penn Presbyterian, Philadelphia, Pennsylvania
  - Addiction Medicine Services, Pittsburgh, Pennsylvania
  - Morris Village/LRADAC, Columbia, South Carolina
  - Nexus Recovery Services, Dallas, Texas

REFERENCES:
- [Background] Winhusen T, Brady KT, Stitzer M, Woody G, Lindblad R, Kropp F, Brigham G, Liu D, Sparenborg S, Sharma G, Vanveldhuisen P, Adinoff B, Somoza E. Evaluation of buspirone for relapse-prevention in adults with cocaine dependence: an efficacy trial conducted in the real world. Contemp Clin Trials. 2012 Sep;33(5):993-1002. doi: 10.1016/j.cct.2012.05.003. Epub 2012 May 19. PMID 22613054
- [Derived] Winhusen TM, Kropp F, Lindblad R, Douaihy A, Haynes L, Hodgkins C, Chartier K, Kampman KM, Sharma G, Lewis DF, VanVeldhuisen P, Theobald J, May J, Brigham GS. Multisite, randomized, double-blind, placebo-controlled pilot clinical trial to evaluate the efficacy of buspirone as a relapse-prevention treatment for cocaine dependence. J Clin Psychiatry. 2014 Jul;75(7):757-64. doi: 10.4088/JCP.13m08862. PMID 24911028

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Buspirone Plus TAU | Placebo Plus TAU
Started | 35 | 27
Completed | 33 | 25
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics of all randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Buspirone Plus TAU | Placebo Plus TAU | Total
Number analyzed (Participants) | 35 | 27 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 27 | 62
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 24 | 15 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 35 | 27 | 62
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 26 | 19 | 45
  White | 8 | 6 | 14
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 35 | 27 | 62

OUTCOME MEASURES:

1. Primary Outcome: Maximum Days of Continuous Cocaine Abstinence
Description: The primary outcome measure selected for the present two-stage protocol is the maximum days of continuous cocaine abstinence during study weeks 4-15. The Timeline Follow-back (TLFB) procedure (Sobell and Sobell, 1992; Fals-Stewart, 2000) will be used to assess the participants' self-reported use of substances for each day of the study. A rapid UDS system that screens for drugs of abuse will be used to analyze the urine samples.
Time Frame: study week 16
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Buspirone Plus TAU | Placebo Plus TAU
Number analyzed (Participants) | 35 | 27
Days | 42.9 (30.83) | 46.6 (31.03)

2. Secondary Outcome: Cocaine-use Days
Description: Cocaine use days during days 22-105 as assessed by UDS and self-report combined with no imputation
Time Frame: study week 16
Population: All randomized participants
Measure: Number; unit: proportion of cocaine use days
Arm/Group | Buspirone Plus TAU | Placebo Plus TAU
Number analyzed (Participants) | 35 | 27
proportion of cocaine use days | 0.153 | 0.134

ADVERSE EVENTS:
Time Frame: Between the first dose of study drug and the last dose of study drug plus 7 days, for up to 16 weeks
Arm/Group | Buspirone Plus TAU | Placebo Plus TAU
Serious Adverse Events (participants affected / at risk) | 3/35 | 0/27
Other Adverse Events (participants affected / at risk) | 18/35 | 11/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buspirone Plus TAU (N=35) | Placebo Plus TAU (N=27)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buspirone Plus TAU (N=35) | Placebo Plus TAU (N=27)
Dizziness (Nervous system disorders) | 15 (18) | 1 (1)
Headache (Nervous system disorders) | 8 (8) | 7 (8)
Somnolence (Nervous system disorders) | 3 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 8 (8) | 4 (6)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 8 (11) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (3) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 2 (2)
Weight increased (Investigations) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No